CLINICAL TRIAL: NCT05130983
Title: A Phase I Study of ExoFlo, an Ex Vivo Culture-expanded Adult Allogeneic Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicle Isolate Product, for the Treatment of Medically Refractory Crohn's Disease
Brief Title: Study of ExoFlo for the Treatment of Medically Refractory Crohn's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment challenges.
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB-EF-CD-01
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases
Keywords: ExoFlo; Inflammatory Bowel Diseases; Crohn's Disease; Extracelluar Vesicle
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 15ml at Day 0, 2, 4, 30 ml at Week 2, Week 6, and every 4 weeks after to week 46 (Experimental): IV administration of 15 mL study agent at Day 0, Day 2, Day 4 and 30 mL at Week 2, Week 6 and every 4 weeks thereafter to week 46 (total # doses = 15).
  Interventions: Biological: ExoFlo

INTERVENTIONS:
Biological: ExoFlo — Intravenous administration of bone marrow mesenchymal stem cell derived extracellular vesicles

SUMMARY:
Protocol Summary

* Title: A Phase I study of ExoFlo, an ex vivo culture-expanded adult allogeneic bone marrow mesenchymal stem cell derived extracellular vesicle isolate product, for the treatment of medically refractory Crohn's disease.
* Short Title: ExoFlo for Crohn's Disease
* Phase: 1
* Methodology: Open label
* Study Duration: 24 months
* Subject Participation: 58 weeks
* Single or Multi-Site: Multi-Site

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the feasibility of intravenous ExoFlo in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies.
* To evaluate the safety of intravenous ExoFlo in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies.

Secondary Objectives:

* To evaluate the efficacy of intravenous ExoFlo in inducing clinical remission in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies.
* To evaluate the efficacy of intravenous ExoFlo in inducing clinical response in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies.
* To evaluate the efficacy of intravenous ExoFlo in improving disease-specific health-related quality of life.
* To evaluate the pharmacokinetics and pharmacodynamics of ExoFlo therapy, including changes in C-reactive protein (CRP) and fecal calprotectin.

Number of Subjects: 10

Diagnosis and Main Inclusion Criteria: Subjects must have colitis, ileitis, or ileocolitis previously confirmed at any time in the past by radiography, histology, and/or endoscopy, and must allow a ≥ 8-week washout for prior monoclonal antibody therapy.

Study Product, Dose, Route, Regimen:

IV administration of 15 mL study agent at Day 0, Day 2, Day 4 and 30 mL at Week 2, Week 6 and every 4 weeks thereafter to week 46 (n=10), (total # doses =15)

Statistical Methodology: This is a safety study with exploratory assessment of efficacy. The study has insufficient power to confirm efficacy. All assessments of efficacy will be exploratory for the purpose of hypothesis-generation in larger sample sizes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-75 years of age
2. Crohn's colitis of at least 6 months duration with medically refractory symptoms who has failed one monoclonal antibody therapy (failed to have improvement of disease while receiving at least one monoclonal antibody for 8 weeks duration prior to enrollment, including, but not limited to, Infliximab, Adalimumab, Certolizumab, Golimumab, Vedolizumab, Ustekinumab and Tofacitinib), or is intolerant, or has a contraindication to monoclonal antibody therapy with a next step of subtotal colectomy or escalation in medical management
3. Patient with medically refractory Crohn's disease as defined by a CDAI score ≥150 and/or SES-CD score ≥ 3
4. Exposure to corticosteroids, 5-ASA drugs, thiopurines, methotrexate, anti-TNF therapy, anti-integrin and anti-interleukin in the past are permitted but a washout period of 8 weeks for any monoclonal antibody is necessary.

   1. If receiving conventional immunomodulators (ie, AZA, 6-MP, or MTX), must have been taking them for ≥12 weeks, and on a stable dose for at least 4 weeks prior to receiving the first dose of the study drug.
   2. If AZA, 6-MP, or MTX has been recently discontinued, it must have been stopped for at least 4 weeks prior to receiving the first dose of study drug.
   3. If receiving oral 5-ASA compounds, the dose must have been stable for at least 4 weeks. If receiving oral corticosteroids, the dose must be ≤20 mg/day prednisone or its equivalent and must have been stable for at least 4 weeks prior to receiving the first dose of study drug.
   4. If receiving budesonide, the dose must have been stable for at least 2 weeks prior to receiving the first dose of study drug.
   5. If oral 5-ASA compounds or oral corticosteroids (including budesonide) have been recently discontinued, they must have been stopped for at least 2 weeks prior to receiving the first dose of study drug.
5. The following medications/therapies must have been discontinued before first administration of study agent:

   1. TNF-antagonist therapy (e.g., infliximab, etanercept, certolizumab, adalimumab, golimumab), vedolizumab, ustekinumab for at least 8 weeks.
   2. Cyclosporine, tacrolimus, or sirolimus, for at least 4 weeks.
   3. 6-thioguanine (6-TG) must have been discontinued for at least 4 weeks.
   4. Rectal corticosteroids (i.e., corticosteroids [including budesonide] administered to the rectum or sigmoid colon via foam or enema or suppository) for at least 2 weeks.
   5. Rectal 5-ASA compounds (i.e., 5-ASAs administered to the rectum or sigmoid colon via foam or enema or suppository) for at least 2 weeks.
   6. Parenteral corticosteroids for at least 2 weeks.
   7. Total parenteral nutrition (TPN) for at least 2 weeks.
   8. Antibiotics for the treatment of CD (e.g., ciprofloxacin, metronidazole, or rifaximin) for at least 2 weeks.
6. No colonic dysplasia and malignancy as ruled out by colonoscopy within 90 days of first ExoFlo delivery
7. Ability to comply with protocol
8. Competent and able to provide written informed consent
9. Stated willingness to comply with all study procedures and availability for the duration of the study
10. If patient is of reproductive capacity, willing to use adequate birth control measures while they are in the study

Exclusion Criteria:

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of ExoFlo: e.g., myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Patients with confirmed HIV, Hepatitis B, or Hepatitis C infections
4. Abnormal AST or ALT at screening defined as AST >100 or ALT > 100
5. Abnormal basic laboratory values with the following cut-offs:

   1. Alkaline phosphate >200
   2. WBC >13
   3. Hemoglobin <7
   4. Platelets <50 or > 1 million
   5. eGFR < 60
   6. HbA1C > 8%
6. Subjects with abnormal coagulation studies:

   1. Prothrombin time (PT) > 1.5 times the upper limits of normal
   2. Partial thromboplastin time (aPTT) > 1.5 times the upper limits of normal
   3. International normalized ratio (INR) > 1.5 times the upper limits of normal
7. Subjects with hyperbilirubinemia and evidence of liver disease as defined by AST > 100 or ALT > 100 or PT > 1.5 times the upper limits or normal or PT/INR > 1.5 time the upper limits of normal.
8. Subjects with abnormal vital signs prior to first ExoFlo delivery as defined by:

   1. Systolic blood pressure >160 or <90 mmHg
   2. Diastolic blood pressure >90 or <60 mmHg
   3. Pulse <60 or >105 bpm
   4. Respiratory Rate <9 and >25 breaths per minute
   5. Temperature: >100.4 degrees Fahrenheit
   6. SpO2: <92%
9. History of cancer including melanoma (with the exception of localized skin cancers) within 5 years of study enrollment
10. Investigational drug within one year of study enrollment
11. Pregnant or breast feeding.
12. If patient is of reproductive capacity, unwilling to use adequate birth control measures while they are in the study
13. Fulminant colitis requiring emergency surgery
14. Concurrent active clostridium difficile infection of the colon
15. Concurrent CMV infection of the colon via colonic biopsy with CMV stain taken within 90 days
16. Evidence of colonic perforation
17. Massive hemorrhage from the colon requiring emergent surgery in the 6 months prior to screening.
18. Ulcerative colitis or indeterminate colitis
19. Microscopic, ischemic or infectious colitis
20. Neoplasia of the colon on preoperative biopsy
21. Presence of an ostomy
22. Three or more prior small bowel resections
23. Previous colonic resection
24. Colonic stricture that unable to pass an adult colonoscope
25. Active or latent tuberculosis
26. Unable to wean off corticosteroids
27. Patients with primary sclerosing cholangitis
28. Patients with history of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 90 days of study entry
29. Patients with known allergy to local anesthetics
30. Patients taking anticoagulant medications (e.g. warfarin, heparin) or clopidogrel (Plavix) to reduce the risk of bleeding/ hemarthrosis
31. Individuals with previously diagnosed, known inherited or acquired hypercoagulable states.
32. Electrocardiogram demonstrating cardiac arrhythmia, except for sinus tachycardia within the predefined limit of no greater than 105 bpm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Safety of intravenous ExoFlo in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies. | 58 Weeks
  Safety will be defined as lack of serious adverse events or adverse advents related to treatment with the study therapeutic.
Feasibility of intravenous ExoFlo in subjects with medically refractory Crohn's disease who have failed, or are intolerant, or have a contraindication to one or more monoclonal antibodies. | 58 Weeks
  The study will not be considered feasible if more than three subjects are not capable of receiving the ExoFlo based on ability to release or deliver the cells. If a subject misses any single dose of ExoFlo, they will be withdrawn and not replaced.

SECONDARY OUTCOMES:
To evaluate the efficacy of intravenous ExoFlo in inducing clinical remission at week 6 and week 46. | Week 6 and Week 46
  Efficacy in inducing clinical remission will be evaluated as a reduction from baseline in the CDAI score of >100 points.
To evaluate the efficacy of intravenous ExoFlo in inducing clinical response at week 6 and week 46. | Week 6 and Week 46
  Efficacy in inducing clinical response will be evaluated as ≥70-point decrease in CDAI score from baseline (Week 0).
To evaluate endoscopic remission and endoscopic response. | 58 Weeks
  Endoscopic remission as measured by an SES-CD score of 0 to 2, and endoscopic response as defined by a 50% reduction in the SES-CD score from baseline.
To evaluate the efficacy of intravenous ExoFlo in improving disease-specific health-related quality of life. | 58 Weeks
  Efficacy will be evaluated as:
  * Improvement on the 36 Item Short Form Health Survey (SF-36)
  * Improvement on the EuroQol 5 Dimensions Survey (EQ-5D)
To evaluate the pharmacokinetics and pharmacodynamics of ExoFlo therapy, including changes in C-reactive protein (CRP) and fecal calprotectin. | 58 Weeks
  Evaluated as:
  Measuring changes in C-reactive protein (CRP) and fecal calprotectin.
To evaluate treatment failure as defined by disease worsening, need for rescue medications or surgical intervention for treatment of CD, or study drug-related adverse event leading to discontinuation from the study. | 58 Weeks
  Evaluated as:
  Number of subjects with disease worsening, needing rescue medications or surgical intervention for treatment of CD, or study drug-related adverse events leading to discontinuation of study.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC
Locations (2):
- United States (2):
  - Direct Biologics Investigational Site, Los Angeles, California
  - Direct Biologics Investigational Site, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Direct Biologics, LLC — https://directbiologics.com/